CLINICAL TRIAL: NCT01368354
Title: Impact of Community-Led Total Sanitation on the Control of Taenia Solium and Soil Transmitted Helminths in the Eastern Province of Zambia
Brief Title: Taenia Solium Control Case Study in Zambia
Acronym: SANTOSOIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zambia (Other)
Responsible Party: Principal Investigator, Chummy S.Sikasunge, Dr. Chummy Sikalizyo Sikasunge, University of Zambia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICONZ-UNZA
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Cysticercosis; Helminthiasis
Keywords: Community Led Total Sanitation; Open Defecation; Cysticercosis; Soil transmitted helminths; Zambia
MeSH Terms: conditions — Cysticercosis; Helminthiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CLTS Arm (Active Comparator): To induce behavioural changes by confronting the community with their open defecation behaviour. This will lead to voluntary construction and use of latrines and improved hygiene behaviour. CLTS involves facilitating a process to inspire and empower rural communities to stop open defecation and to build and use latrines, without offering external hardware subsidies. Communities are encouraged to appraise and analyse their own sanitation profile, including the extent of open defecation and the spread of faecal-oral contamination.
  Interventions: Behavioral: CLTS
- Control arm (No Intervention)

INTERVENTIONS:
Behavioral: CLTS — CLTS (Community Led Total Sanitation) involves facilitating a process to inspire and empower rural communities to stop open defecation and to build and use latrines, without offering external hardware subsidies. Communities are encouraged to appraise and analyse their own sanitation profile, including the extent of open defecation and the spread of faecal-oral contamination. This approach ignites a sense of disgust and share among the community. The community then collectively realises the impact of its unsanitary practices and this realisation mobilises and initiates collective action to improve the existing sanitation profile.
  Arms: CLTS Arm

SUMMARY:
Summary Diseases due to T. solium and soil transmitted helminths (STHs) are of cosmopolitan distribution and strongly linked with poor sanitation and poverty. These infections are to a great extent perpetuated by open defecation (OD). Community-Led Total Sanitation (CLTS) is an approach in which people in rural communities are facilitated to do their own appraisal and analysis, come to their own conclusions, and take their own actions. To date no rigorous study has been conducted to evaluate the impact of CLTS on the transmission of taeniasis/cysticercosis or STHs, despite the worldwide acclaim which CLTS has received as an approach to improve sanitation. The overall aim of the study is to contribute to the reduction and subsequent control of T. solium and STH infections through the implementation of CLTS approaches in 1 districts in the Eastern Province of Zambia. By using CLTS it is hypothesised that toilet acquisition and usage will be increased with a resultant reduction in OD which will in turn reduce the transmission of T. solium and STH infections in the district. This will be measured by porcine/human cysticercosis prevalence (serological test) and STH infections in humans (quantitative coprological test).

DETAILED DESCRIPTION:
The study procedure will consist of conducting a pilot study with census to establish the sample frame, shortly followed by a baseline survey during which baseline data on human cysticercosis, porcine cysticercosis (serological test), STH infection prevalence (quantitative coprological test) and anthropometric data (weight, height, arm circumference) will be obtained from the study communities (infected people will receive treatment). The study communities will be subsequently randomly allocated a status of intervention or control community, and this will determine the point at which CLTS will be administered, but all communities will ultimately receive CLTS. CLTS will be conducted in intervention communities for 12 months by UNICEF. A post-intervention survey will follow the 12 month CLTS campaign, and all factors investigated at baseline will be revisited in both intervention and control communities. The compliance of the CLTS approach will also be measured. CLTS will be administered to control communities after the completion of the post-intervention survey. Baseline data will be used to show that the groups are comparable; in the primary analysis the difference between intervention and control at follow up will be analyzed to evaluate the impact of CLTS. If this intervention can be demonstrated to have an impact on the occurrence and burden of sanitation-linked diseases, then this will provide advocacy for such an approach at policy-maker level.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to collaborate
* Accessible by road all year round, even during the wet season
* No current promotion of water, sanitation or hygiene programs
* Rural setting
* Minimum of 10 pig-keeping households (HHs)
* Maximum of 100 HHs

Exclusion Criteria:

* Other ongoing sanitation programmes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1197 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of porcine/human cysticercosis cases (serological test) | One Year
  Blood samples will be collected from humans and pigs before and after intervention in both study arms. Sera will be tested for presence of circulating cysticercus antigens by a monoclonal antibody based antigen capturing ELISA. Test result above cut-off is positive.

SECONDARY OUTCOMES:
Number of STH cases in humans | 1 year
  All willing participants will be faecal sampled before and after intervention in both study arm. Samples will be analysed by a quantitative coprological test (Mc Master method) for measuring presence and levels of soil transmitted helminths (ascaris, trichuris and hookworm). An EPG (eggs per gram) count will be determined for each worm species. It is anticipated that CLTS will have an impact (reduction) on faecal contamination of the environment thereby reducing transmission of STH

CONTACTS AND LOCATIONS:
Overall Officials: Chummy Sikasunge, PhD, Principal Investigator — University of Zambia; Evans K. Mwape, MSc, Principal Investigator — University of Zambia; Sarah Gabriel, PhD, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium; Pierre Dorny, PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium; Giveson Zulu, PhD, Principal Investigator — UNICEF
Locations (1):
- Katete, Katete District, Eastern Province, Zambia